CLINICAL TRIAL: NCT06758817
Title: The Triad of Nutrition, Intestinal Microbiota and Rheumatoid Arthritis (TASTY)
Acronym: TASTY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lisbon Academic Medical Center - Centro Académico de Medicina de Lisboa (Network)
Collaborators: Gulbenkian Institute for Molecular Medicine (Other)
Responsible Party: Principal Investigator, Ana Lopes, Centro Académico de Medicina de Lisboa, Lisbon Academic Medical Center - Centro Académico de Medicina de Lisboa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASTY; Grant No: 2022.07462 (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia, FCT); Grant No: 101095084 (Other Grant/Funding Number: European Union (ENDOTARGET © Project)); Contract No: 22.00462 (Other Grant/Funding Number: Swiss Secretariat - Education, Research, Innovation (SERI)); Grant No: 101093997 (Other Grant/Funding Number: European Union (GlycanTrigger © Project))
Record Dates: First submitted 2024-12-12; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Diet Interventions
Keywords: Diet Interventions; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Block randomization was performed through an online software, and patients are being allocated into the intervention (MedDiet+) or control groups. Due to the nature of the trial, the participants and the dietitians responsible for implementing the study are not blinded. However, the clinicians evaluating the clinical outcome measures (disease activity score in 28 joints and the doppler ultrasound score in 32 joints) and the researchers performing the laboratory tests are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MedDiet+ intervention (Experimental): The 12-week nutritional intervention includes a personalized dietary plan based on the MedDiet+ pattern, educational resources, food basket deliveries, and clinical culinary workshops, all developed and monitored weekly by registered dietitians. The nutritional plan includes the food portions of each food group in agreement with the MedDiet recommendations for the adult population, complemented with fermented foods including kefir (provided for daily consumption) and kombucha (provided for consumption 2x/week).
  Interventions: Other: MedDiet+ intervention
- General dietary recommendations (Active Comparator): This group receives a flyer with general recommendations on a healthy diet based on the Portuguese brief guidance for healthy eating in primary health care at baseline
  Interventions: Other: General dietary recommendations

INTERVENTIONS:
Other: MedDiet+ intervention — Study arm will consume a Mediterranean like style diet enriched in fermented foods for 12 weeks
  Arms: MedDiet+ intervention
Other: General dietary recommendations — Study arm will be given general healthy eating advice at baseline.
  Arms: General dietary recommendations

SUMMARY:
The main goal of this trial is to investigate whether a dietary intervention based on a typical Mediterranean Diet enriched with fermented foods (MedDiet+) can impact gut microbiota and RA-related outcomes.

DETAILED DESCRIPTION:
100 RA patients will be recruited at ULS Santa Maria in Lisbon, Portugal, and randomly assigned to either the intervention (MedDiet+) or the control group. The 12-week nutritional intervention will include a personalized dietary plan based on the MedDiet+ pattern, educational resources, food basket deliveries, and clinical culinary workshops, all developed and monitored weekly by registered dietitians. The control group will receive general recommendations for a healthy diet at baseline. The intervention's effects will be assessed by evaluating disease activity, functional status, quality of life, intestinal permeability, endotoxemia, inflammatory biomarkers, intestinal and oral microbiota, serum proteomics, and serum glycome profile characterisation.

ELIGIBILITY:
Inclusion Criteria:

* RA patients (ACR/EULAR2010 criteria)
* Age >18-years
* Disease duration >1-year
* Active disease (DAS28 > 2.6units)
* On stable medication for 12 weeks
* Low/medium MedDiet adherence (PREDIMED<10)
* Willing to comply with study protocol

Exclusion Criteria:

* Prednisolone dose ≥ 7.5 mg/day
* Antibiotic therapy 4-weeks prior to baseline
* Persistent use of NSAID's
* Inflammatory or irritable bowel disease
* Celiac disease
* Chronic diarrhea
* Diabetes
* Other immune-mediated inflammatory diseases besides RA
* Major organ dysfunction
* Cancer diagnosed in the last five years
* Health conditions which may difficult participation (cognitive impairment/psychiatric disease)
* Pregnant or lactating individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DAS28-ESR | 12 weeks
  Disease Activity Score in 28 Joints Calculated with erythrocyte sedimentation rate (DAS28-ESR), higher scores indicate higher disease activity

SECONDARY OUTCOMES:
EULAR Good or Moderate Response | 12 weeks
  Proportion of patients achieving moderate or good response based on European Alliance of Associations for Rheumatology (EULAR) criteria; measured with Disease Activity Score using Erythrocyte Sedimentation Rate) (DAS28-ESR<2.6 (%).
Ultrasound score | 12 weeks
  i. Change in ultrasound score for 32 joints assessed using a 0-3 scale for grey scale and power Doppler, score (0-3) per joint, higher scores indicate worse disease activity.
  ii. Proportion of patients achieving a 10% improvement in the ultrasound joint score (%).
DAS28-CRP | 12 weeks
  Change in Disease Activity Score in 28 joints calculated with C-reactive protein (DAS28-CRP), higher scores indicate worse disease activity.
Quality of life | 12 weeks
  Change in Short Form-36 (SF-36): higher scores indicate better quality of life, score ranging from 0 to 100
Functional status | 12 weeks
  Change in Health Assessment Questionnaire (HAQ): higher scores indicate greater disability, score ranging from 0 to 3
α- and β- diversity of the gut and oral microbiota | 12 weeks
  i. Change in α-diversity: changes in alpha diversity between the different groups using the Chao-1 index, Phylogenetic Diversity index, Simpson index, and Shannon index.
  ii. Change in β-diversity: we will perform Principal Coordinates Analysis (PCoA) using Bray-Curtis dissimilarity, Weighted UniFrac, and Unweighted
Changes in key gut microbial species | 12 weeks
  i. Change in the relative abundance of Lactobacillus/ Limosilactobacillus and Bifidobacterium, relative abundance in percentage. ii. Change in butyrate-producing species, relativ abundance in percentage. iii. Change in H₂S-producing species, relative abundance in percentage.
Intestinal permeability | 12 weeks
  Change in the lactulose/mannitol ratio
Endotoxemia | 12 weeks
  Change in Endotoxemia measured by TLR4 activation in reporter cells
CRP | 12 weeks
  Change in C-reactive protein (CRP, mg/L)
ESR | 12 weeks
  Change in erythrocyte sedimentation rate (ESR, mm/hr)
Faecal calprotectin | 12 weeks
  Change in faecal calprotectin (μg/g)
CD14s | 12 weeks
  Change in serum soluble CD14 (CD14s, ng/mL)
LBP | 12 weeks
  Change in lipopolysaccharide-binding protein (LBP, ng/mL)
IFABP | 12 weeks
  Change in intestinal fatty acids binding protein levels (IFABP, pg/mL)
Lipid Profile | 12 weeks
  i.Change in triglycerides (mg/dL) ii.Change in total cholesterol (mg/dL) iii.Change in high-density lipoprotein cholesterol (HDL, mg/dL) iv.Change in low-density lipoprotein cholesterol (LDL, mg/dL)
Body composition | 4 th, 8 th and 12 th weeks
  Change in body mass index (BMI, kg/m²; weight in kilograms and height in meters will be comined to report BMI in kg/m²)
Anthropometric measurements | 4 th, 8 th and 12 th weeks
  Change in body mass index and waist circumference
Waist circunference | 4 th, 8 th and 12 th weeks
  Change in waist circumference (cm)

OTHER OUTCOMES:
zonulin levels, serum proteomics, and serum glycomics | 12 weeks
  We will also analyse:
  i. Change in zonulin levels (ng/mL). ii. Change in serum proteomics. iii. Change in serum glycomics.

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Sousa Guerreiro, RD PhD, Principal Investigator — Nutrition Lab, Faculty of Medicine, University of Lisbon
Locations (2):
- Portugal (2):
  - Unidade Local de Saude de Santa Maria, Lisbon, Portugal
  - Faculdade Medicina de Lisboa, Lisbon, Portugal

REFERENCES:
- [Derived] Charneca S, Hernando A, Almada-Correia I, Polido-Pereira J, Vieira A, Sousa J, Almeida AS, Motta C, Barreto G, Eklund KK, Alonso-Perez A, Gomez R, Cicci F, Mauro D, Pinho SS, Fonseca JE, Costa-Reis P, Guerreiro CS. TASTY trial: protocol for a study on the triad of nutrition, intestinal microbiota and rheumatoid arthritis. Nutr J. 2025 Apr 7;24(1):52. doi: 10.1186/s12937-025-01089-6. PMID 40189532